CLINICAL TRIAL: NCT04785469
Title: Impact of a Low-load Eccentric Training Program on Peripheral Muscle Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Eccentric Training in Individuals With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Eccentric Training_COPD_FDG
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-03

CONDITIONS: Copd
Keywords: Copd; Pulmonary rehabilitation; Muscle strength; Resistance training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric training group (Experimental)
  Interventions: Other: Low-load eccentric training
- Control group (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Low-load eccentric training — * Aerobic exercise training on a downhill walking treadmill with the following settings: 10% negative incline and constant speed corresponding to 75% of the average speed recorded during the initial 6-Minute walk test.
  * Resistance training: 5 minutes of warm-up on the manual ergometer, then 3 sets for 10 repetitions of the leg extension (performed unilaterally in eccentric phase) with a load of 75% of 1 repetition maximum (concentric) for the first two weeks. The following two weeks, 3 sets for 10 repetitions will be performed on the leg press (performed unilaterally in the eccentric phase) with 75% load of 1 repetition maximum (concentric). In addition, patients will perform 3 upper extremity strengthening exercises (free weights or elastic bands), including 2 sets of 10 repetitions for each exercise.
  Arms: Eccentric training group
Other: Usual care — * Aerobic exercise training using the cycle ergometer at an intensity calculated as follows: 2 minutes with load equal to 20% of maximum load, then 25 minutes with initial load at 50% of maximum load calculated as 103.217 + (30.500xGender) + (-1.613xAge) + [0.002x6-Minute walk work (6MWW)]. [Sex: female = 0; male:1] [6MWW = 6-Minute walk distance x weight in kg].
  * Resistance training: 5 minutes of warm-up on the manual ergometer, then 5 exercises for upper and lower limbs performed with free weights or elastic bands. For the first 2 weeks will be performed 2 sets X 20 repetitions with 1 minute break between sets and a load that allows to perform no more than 20 repetitions. For the following 2 weeks, 3 sets of 10 repetitions x 10 repetitions with 2 min break between sets and a load that allows for no more than 10 repetitions.
  Arms: Control group

SUMMARY:
Skeletal muscle dysfunction as a systemic consequence of chronic obstructive pulmonary disease (COPD) has a major impact on quality of life, health care resource utilization, and mortality of patients with this disease. In fact, a vicious circle of inactivity and disuse is established in the advanced stages of the disease, inducing a progressive decline in exercise tolerance and a loss of muscle mass (especially in locomotor muscles), resulting in the inability of patients to perform even the simplest daily activities.

In this context, the multidisciplinary rehabilitation approach includes not only recovery of exercise capacity but also training aimed at restoring muscle function in patients with COPD. However, there is considerable methodological variability among muscle resistance training programs used in clinical practice with patients with COPD. This is compounded by the need to identify alternative training strategies effective in inducing functional adaptation in skeletal muscle without increasing the degree of dyspnea or fatigue in those symptomatic patients with advanced stages of disease. Among these, eccentric exercise or negative work, i.e. the stretching of the muscle during the active contraction phase, represents a valid alternative to traditional concentric training in various rehabilitation contexts. The main advantages of this training method are: 1) eccentric contraction is able to produce greater forces than isometric and concentric contraction; 2) for the same resistance, eccentric contraction has a lower metabolic cost than concentric contraction. For these reasons, eccentric exercise is a valid method of muscle strengthening in rehabilitation and in particular in those subjects unable to sustain a high cardiorespiratory effort, as in the case of patients with moderate-severe COPD. Previous studies have also shown that eccentric exercise, even at low load, produces results equivalent if not superior to traditional training with respect to some particular characteristics of muscle function such as power and hypertrophy.

However, eccentric training programs for muscle dysfunction recovery in patients with COPD are underused in clinical practice, so far. In contrast, the so called iso-weight eccentric training, more suitable for clinical practice, could also be applied to rehabilitation programs designed for COPD patients.

The aim of this study is therefore to evaluate the reliability and efficacy of a low-load eccentric exercise training program compared to usual care for the improvement of muscle function in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis (GOLD stage: II-III-IV), defined as post-bronchodilator forced expiratory volume in 1s (FEV1)/forced vital capacity < 0.7 and FEV1 < 80% predicted.

Exclusion Criteria:

* Restrictive lung disease, unstable conditions, recent exacerbation, infection, embolism, pneumothorax, thoracic or abdominal surgery (less than 3 months before recruitment).
* Cardiologic conditions like myocardial infarction (less than 6 months before recruitment), heart failure, or severe angina.
* Inability of perform the exercise training (e.g. orthopaedic conditions).
* Incapability to understand the instructions required to carry out the tests and assessments planned.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Maximal muscle strength | Change from baseline up to 4 weeks
  Isometric peak torque of the quadriceps.

SECONDARY OUTCOMES:
Six-minute walk distance | Change from baseline up to 4 weeks
  The distance that an individual can walk on an indoor 30-m flat corridor for a 6-min period.
Mobility function | Change from baseline up to 4 weeks
  The Short Physical Performance Battery (SPPB) is a test made by 3 components (standing balance, 4-m gait speed, and 5-repetitions sit-to-stand) measured by total time and kinematic parameters.
Muscle function | Change from baseline up to 4 weeks
  Measures of muscle accuracy and steadiness intended as the ability to control muscle force performing submaximal contractions during standardized tasks.
Body composition | Change from baseline up to 4 weeks
  Fat-free mass Index (FFM; calculated as the sum of lean mass and bone mineral mass)
Airways resistance | Change from baseline up to 4 weeks
  Measure of airway Resistance [Rrs (cmH2O/L/s)]
Airways reactance | Change from baseline up to 4 weeks
  Measure of airway Reactance [Xrs (cmH2O/L/s)]

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

REFERENCES:
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Barreiro E, Gea J. Respiratory and Limb Muscle Dysfunction in COPD. COPD. 2015 Aug;12(4):413-26. doi: 10.3109/15412555.2014.974737. PMID 25438125
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Bourbeau J, De Sousa Sena R, Taivassalo T, Richard R, Jensen D, Baril J, Rocha Vieira DS, Perrault H. Eccentric versus conventional cycle training to improve muscle strength in advanced COPD: A randomized clinical trial. Respir Physiol Neurobiol. 2020 May;276:103414. doi: 10.1016/j.resp.2020.103414. Epub 2020 Feb 9. PMID 32050099
- [Background] Roig M, Shadgan B, Reid WD. Eccentric exercise in patients with chronic health conditions: a systematic review. Physiother Can. 2008 Spring;60(2):146-60. doi: 10.3138/physio.60.2.146. Epub 2008 Oct 10. PMID 20145778
- [Background] LaStayo P, Marcus R, Dibble L, Frajacomo F, Lindstedt S. Eccentric exercise in rehabilitation: safety, feasibility, and application. J Appl Physiol (1985). 2014 Jun 1;116(11):1426-34. doi: 10.1152/japplphysiol.00008.2013. Epub 2013 Jul 3. PMID 23823152
- [Background] Ellis R, Shields N, Lim K, Dodd KJ. Eccentric exercise in adults with cardiorespiratory disease: a systematic review. Clin Rehabil. 2015 Dec;29(12):1178-97. doi: 10.1177/0269215515574783. Epub 2015 Mar 10. PMID 25758944
- [Background] Raj IS, Bird SR, Westfold BA, Shield AJ. Effects of eccentrically biased versus conventional weight training in older adults. Med Sci Sports Exerc. 2012 Jun;44(6):1167-76. doi: 10.1249/MSS.0b013e3182442ecd. PMID 22143107
- [Background] Douglas J, Pearson S, Ross A, McGuigan M. Chronic Adaptations to Eccentric Training: A Systematic Review. Sports Med. 2017 May;47(5):917-941. doi: 10.1007/s40279-016-0628-4. PMID 27647157
- [Background] Franchi MV, Maffiuletti NA. Distinct modalities of eccentric exercise: different recipes, not the same dish. J Appl Physiol (1985). 2019 Sep 1;127(3):881-883. doi: 10.1152/japplphysiol.00093.2019. Epub 2019 May 9. No abstract available. PMID 31070957
- [Background] Luxton N, Alison JA, Wu J, Mackey MG. Relationship between field walking tests and incremental cycle ergometry in COPD. Respirology. 2008 Nov;13(6):856-62. doi: 10.1111/j.1440-1843.2008.01355.x. PMID 18811884
- [Background] Medina-Mirapeix F, Bernabeu-Mora R, Llamazares-Herran E, Sanchez-Martinez MP, Garcia-Vidal JA, Escolar-Reina P. Interobserver Reliability of Peripheral Muscle Strength Tests and Short Physical Performance Battery in Patients With Chronic Obstructive Pulmonary Disease: A Prospective Observational Study. Arch Phys Med Rehabil. 2016 Nov;97(11):2002-2005. doi: 10.1016/j.apmr.2016.05.004. Epub 2016 May 30. PMID 27255806
- [Background] Franssen FM, Rutten EP, Groenen MT, Vanfleteren LE, Wouters EF, Spruit MA. New reference values for body composition by bioelectrical impedance analysis in the general population: results from the UK Biobank. J Am Med Dir Assoc. 2014 Jun;15(6):448.e1-6. doi: 10.1016/j.jamda.2014.03.012. Epub 2014 Apr 20. PMID 24755478
- [Background] Tracy BL, Enoka RM. Older adults are less steady during submaximal isometric contractions with the knee extensor muscles. J Appl Physiol (1985). 2002 Mar;92(3):1004-12. doi: 10.1152/japplphysiol.00954.2001. PMID 11842033
- [Background] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Derived] Pancera S, Lopomo NF, Porta R, Sanniti A, Buraschi R, Bianchi LNC. Effects of Combined Endurance and Resistance Eccentric Training on Muscle Function and Functional Performance in Patients With Chronic Obstructive Pulmonary Disease: Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Mar;105(3):470-479. doi: 10.1016/j.apmr.2023.09.004. Epub 2023 Sep 15. PMID 37716519